CLINICAL TRIAL: NCT06160414
Title: A Phase 1 Study to Evaluate the Potential Drug Interactions Between ALXN2080 and Rosuvastatin and Metformin in Healthy Adult Participants
Brief Title: A Study to Investigate the Potential Drug Interactions Between ALXN2080 and Rosuvastatin and Metformin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7420C00002
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: rosuvastatin; ALXN2080; metformin
MeSH Terms: interventions — Metformin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): On Day 1, all participants will receive a single oral dose (fasted) of Metformin followed by a single oral dose (fasted) of Rosuvastatin on Day 3.
  Interventions: Drug: Metformin; Drug: Rosuvastatin
- Cohort 2 (Experimental): All participants will receive ALXN2080 twice daily (BID) on Day 1 to Day 11. On the morning of Day 6, participants will be given a single dose of Metformin co-administered with the morning dose of ALXN2080. On the morning of Day 8, participants will be given a single dose of Rosuvastatin co-administered with the morning dose of ALXN2080.
  Interventions: Drug: Metformin; Drug: Rosuvastatin; Drug: ALXN2080

INTERVENTIONS:
Drug: Metformin — Participants will receive Metformin orally, after fasting.
Drug: Rosuvastatin — Participants will receive Rosuvastatin orally, after fasting.
Drug: ALXN2080 — Participants will receive ALXN2080 orally, after fasting.
  Arms: Cohort 2

SUMMARY:
The primary objectives of this study are to determine the effect of multiple doses of ALXN2080 on the single-dose PK of rosuvastatin and to determine the effect of multiple doses of ALXN2080 on the single-dose PK of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, triplicate 12-lead ECG, screening clinical laboratory profiles (hematology, clinical chemistry, coagulation, and urinalysis), as deemed by the Investigator or designee.
* Body Mass Index (BMI) within the range of 18.0 to 32.0 kg/m2 (inclusive) and a minimum body weight of 50.0 kg at screening.
* Female participants of childbearing potential and male participants must follow protocol-specified contraception guidance.

Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological or other disorders.
* History of meningococcal infection.
* History of additional risk factors for Torsades de Pointes (eg, heart failure, hypokalemia, family history of Long QT syndrome).
* History of clinically significant hypersensitivity or idiosyncratic reaction to the study intervention or related compounds.
* History of unexplained, recurrent infection, or infection requiring treatment with systemic antibiotics within 14 days prior to Period 1 Day 1.
* History of significant multiple and/or severe allergies (hay fever is allowed unless it is active), including significant hypersensitivity reactions to commonly used antibacterial agents, including beta-lactams, penicillin, amoxicillin, aminopenicillin, fluoroquinolones (specifically including ciprofloxacin), cephalosporins, and carbapenems, which in the opinion of the Investigator would make it difficult to provide empiric antibiotic therapy or treat an active infection.
* Diseases or conditions or previous procedures known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within 5 years prior to screening, with the exception of nonmelanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
* Known hepatic or biliary abnormalities (including participants with Gilberts syndrome).
* Participants with a history of cholecystectomy or gall stones.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Rosuvastatin | Day 3 up to Day 12
Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Rosuvastatin | Day 3 up to Day 12
Cmax of Metformin | Day 1 up to Day 9
AUC0-inf of Metformin | Day 1 up to Day 9

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Baseline up to Day 29
Cmax of ALXN2080 | Day 1 up to Day 18
Area Under the Plasma Concentration Versus Time Curve for the Defined Interval Between Doses AUC(tau) of ALXN2080 | Day 1 up to Day 18

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR